CLINICAL TRIAL: NCT00002488
Title: INTENSIFICATION WITH HIGH DOSE CYCLOPHOSPHAMIDE, ETOPOSIDE, AND CISPLATIN FOR INTERMEDIATE OR HIGH GRADE LYMPHOMA PATIENTS WHO FAILED PRIMARY COMBINATION CHEMOTHERAPY
Brief Title: Combination Chemotherapy in Treating Patients With Intermediate-Grade or High-Grade Non-Hodgkin's Lymphoma Who Have Not Responded to Anthracycline-Containing Combination Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Regional Cancer Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077375; CAN-OTT-9106; NCI-V92-0013
Record Dates: First submitted 1999-11-01; First posted 2004-08-30 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2000-04

CONDITIONS: Lymphoma
Keywords: recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Cisplatin; Cyclophosphamide; Etoposide

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: etoposide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy consisting of cyclophosphamide, etoposide, and cisplatin in treating patients with intermediate or high-grade non-Hodgkin's lymphoma who have relapsed following or are resistant to anthracycline-containing primary combination chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of high-dose cyclophosphamide/etoposide/cisplatin in patients with intermediate- or high-grade non-Hodgkin's lymphoma who have failed primary combination chemotherapy but still respond to conventional-dose DHAP (dexamethasone/cytarabine/cisplatin) and are not candidates for bone marrow transplantation. II. Determine the toxicity of the intensification chemotherapy regimen in this group of patients.

OUTLINE: Nonrandomized study. 3-Drug Combination Chemotherapy. CVP: Cyclophosphamide, CTX, NSC-26271; Etoposide, VP-16, NSC-141540; Cisplatin, CDDP, NSC-119875.

PROJECTED ACCRUAL: If at least 1 CR is seen in the first 6 patients, an estimated maximum of 20 patients will be enrolled. If 3 or more of the first 10 patients (or 25% of the study population thereafter) die within the first 35 days of treatment from causes unrelated to tumor progression, the study will be terminated.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed intermediate- or high-grade non- Hodgkin's lymphoma of the following histologies: Follicular, predominantly large cell Diffuse small cleaved cell Diffuse mixed, small and large cell Diffuse large cell Large cell, immunoblastic Lymphoblastic Small noncleaved cell Disease has relapsed following or is resistant to primary anthracycline-containing combination chemotherapy Objective response to salvage DHAP chemotherapy required Ineligible for bone marrow transplantation

PATIENT CHARACTERISTICS: Age: 18 to 64 Performance status: Zubrod 0 or 1 Hematopoietic: ANC at least 1,500 Platelets at least 140,000 Hb at least 10 g/dl Hepatic: Bilirubin less than 1.5 mg/dl (26 micromoles/liter) SGOT less than 4 x normal Renal: Creatinine less than 1.5 mg/dl (133 micromoles/liter) Cardiovascular: LVEF greater than 50% No life-threatening arrhythmia by EKG No uncontrolled hypertension Pulmonary: FEV, FVC, and DLCO greater than 50% of predicted Other: No uncontrolled diabetes No other uncontrolled medical condition No history of second malignancy except: Nonmelanomatous skin cancer Carcinoma in situ Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior anthracycline-containing combination chemotherapy required Prior salvage DHAP chemotherapy required Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1991-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C. Yau, MD, Study Chair — Ottawa Regional Cancer Centre
Locations (2):
- Canada (2):
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario